CLINICAL TRIAL: NCT00803101
Title: An Open-label, Randomized, Multicenter Phase IIIb Study to Assess the Efficacy, Safety and Tolerance of BERIPLEX® P/N Compared With Plasma for Rapid Reversal of Coagulopathy Induced by Vitamin K Antagonists in Subjects Requiring an Urgent Surgical Procedure
Brief Title: An Open-label, Randomized, Multicenter Phase IIIb Study to Assess the Efficacy, Safety and Tolerance of BERIPLEX® P/N (Kcentra) Compared With Plasma for Rapid Reversal of Coagulopathy Induced by Vitamin K Antagonists in Subjects Requiring an Urgent Surgical Procedure
Acronym: BE1116_3003
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE1116_3003; 1474 (Other: CSL Behring); 2007-007862-39 (EudraCT Number)
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2014-03

CONDITIONS: Reversal of Coagulopathy
Keywords: Anticoagulant reversal; Prothrombin Complex Concentrate; Coagulopathy; Coumarin derivatives; Emergency surgery; Invasive procedures; Vitamin K; Reversal of coagulopathy induced by coumarin derivatives; Kcentra
MeSH Terms: conditions — Hemophilia B; Hemostatic Disorders

ARMS (2):
- Beriplex® P/N (Experimental)
  Interventions: Biological: Beriplex® P/N (Kcentra)
- Fresh frozen plasma (Active Comparator)
  Interventions: Biological: Fresh frozen plasma

INTERVENTIONS:
Biological: Beriplex® P/N (Kcentra) — Intravenous infusion, dosage depending on baseline INR, amount of coagulation factor IX and body-weight.
  Other Names: Kcentra
  Arms: Beriplex® P/N
Biological: Fresh frozen plasma — Intravenous infusion, dosage depending on baseline INR and body weight
  Arms: Fresh frozen plasma

SUMMARY:
The purpose of this study is to evaluate efficacy, safety and tolerance of Beriplex® P/N (Kcentra) compared with plasma in regard to rapid reversal of coagulopathy induced by vitamin K antagonists in subjects who require immediate correction of international normalized ratio (INR) because of emergency surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects greater than or equal to 18 years,
* Subjects currently on oral vitamin K antagonist (VKA) therapy,
* An urgent surgical procedure is required within 24 hours of the start of investigational medicinal product (IMP),
* Due to the nature of the procedure, withdrawal of oral VKA therapy and infusion of plasma are also indicated to reverse the VKA effect,
* INR greater than or equal to 2 within 3 hours before start of IMP,
* Informed consent has been obtained.

Exclusion Criteria:

* Subjects requiring urgent surgical procedures where according to the surgeon's clinical judgment, an accurate estimate of blood loss is not possible (e.g., ruptured aneurysm),
* Subjects for whom administration of intravenous vitamin K and vitamin K antagonists withdrawal alone can adequately correct the subject's coagulopathy before initiation of the urgent surgical procedure,
* Administration of intravenous vitamin K more than 3 hours or administration of oral vitamin K more than 6 hours prior to infusion of IMP,
* Subjects in whom lowering INR within normal range may present an unacceptable risk for a thromboembolic complication where the INR goal is to lower but not normalize the INR because of risk of a procedure-associated stroke,
* Subjects, who despite medical management that includes close monitoring and diuretics, may not, by investigator assessment, tolerate the total volume of IMP required by the protocol,
* Expected need for additional non-study blood products before infusion of IMP (Note: Administration of packed red blood cells is not an exclusion criterion),
* Expected need for platelet transfusions or desmopressin before Day 10,
* Acute trauma for which reversal of vitamin K antagonists alone would not be expected to control or resolve an acute bleeding complication and/or control the acute bleeding event,
* Unfractionated or low molecular weight heparin use within 24 hours before randomization or potential need before completion of the procedure,
* History of thromboembolic event, myocardial infarction, unstable angina pectoris, critical aortic stenosis, cerebral vascular accident, transient ischemic attack, severe peripheral vascular disease, disseminated intravascular coagulation within 3 months of enrollment,
* Reversal of VKA therapy alone may not resolve the coagulopathy (eg, receiving a potent anti-platelet agent, i.e., clopidogrel or prasugrel, or advanced liver disease),
* Known history of antiphospholipid antibody syndrome or lupus anticoagulant antibodies,
* Suspected or confirmed serious viral or bacterial infection, e.g., meningitis, or sepsis at time of enrollment,
* Administration of whole blood, plasma, plasma fractions or platelets within 2 weeks prior to inclusion into the study (Note: Administration of packed red blood cells is not an exclusion criterion),
* Pre-existing progressive fatal disease with a life expectancy of less than 2 months,
* Known inhibitors to coagulation factors II, VII, IX, or X; or hereditary protein C or protein S deficiency; or heparin-induced, type II thrombocytopenia,
* Treatment with any other investigational medicinal product within 30 days prior to inclusion into the study,
* Presence or history of hypersensitivity to components of the study medication,
* Pregnant or breast-feeding women,
* Prior inclusion in this study or any other CSL Behring sponsored Beriplex study,
* For subjects with intracranial hemorrhage with:

  * Glasgow Coma Score <10 (see Appendix 8)
  * Modified Rankin Score > 3 prior to ICH (see Appendix 9)
  * Intracerebral hemorrhage
  * Epidural hematomas
  * Infratentorial hemorrhage
  * Subarachnoid hemorrhage (SAH) subjects with a Hunt and Hess Scale >2
  * Subdural hematomas that:

    * are judged to be an acute subdural hematoma (based on neurosurgeon review)
    * have a concurrent SAH or parenchymal contusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2009-02; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (30):
- United States (16):
  - Study Site, Newark, Delaware
  - Study site, Lexington, Kentucky
  - Study Site, Boston, Massachusetts
  - Study Site, Duluth, Minnesota
  - Study Site, Minneapolis, Minnesota
  - Study Site, Albuquerque, New Mexico
  - Study Site, Rochester, New York
  - Study Site, Winston-Salem, North Carolina
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, West Reading, Pennsylvania
  - Study Site, Wilkes-Barre, Pennsylvania
  - Study Site, Memphis, Tennessee
  - Study Site, Austin, Texas
  - Study site, Bryan, Texas
  - Study Site, El Paso, Texas
  - Study Site, Houston, Texas
- Belarus (2):
  - Study Site 1, Minsk
  - Study Site 2, Minsk
- Bulgaria (3):
  - Study Site, Rousse
  - Study Site 4, Sofia
  - Study Site, Varna
- Lebanon (2):
  - Study Site, Beirut
  - Study Site, Saida
- Study Site, Timișoara, Romania
- Russia (6):
  - Study Site 2, Barnaul
  - Study Site, Kazan'
  - Study Site 1, Moscow
  - Study Site 2, Moscow
  - Study Site, Novosibirsk
  - Study Site, Saint Petersburg

REFERENCES:
- [Result] Goldstein JN, Refaai MA, Milling TJ Jr, Lewis B, Goldberg-Alberts R, Hug BA, Sarode R. Four-factor prothrombin complex concentrate versus plasma for rapid vitamin K antagonist reversal in patients needing urgent surgical or invasive interventions: a phase 3b, open-label, non-inferiority, randomised trial. Lancet. 2015 May 23;385(9982):2077-87. doi: 10.1016/S0140-6736(14)61685-8. Epub 2015 Feb 27. PMID 25728933
- [Derived] Refaai MA, Goldstein JN, Lee ML, Durn BL, Milling TJ Jr, Sarode R. Increased risk of volume overload with plasma compared with four-factor prothrombin complex concentrate for urgent vitamin K antagonist reversal. Transfusion. 2015 Nov;55(11):2722-9. doi: 10.1111/trf.13191. Epub 2015 Jul 1. PMID 26135740

RESULTS

PARTICIPANT FLOW:
Groups:
- Beriplex® P/N: Beriplex® P/N: Intravenous infusion, dosage depending on baseline international normalized ratio (INR), amount of coagulation factor IX and body-weight.
Period: Overall Study
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Started | 88 | 88
Completed | 70 | 66
Not Completed | 18 | 22
Not completed — Death / Serious Adverse Event | 4 | 6
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 7
Not completed — Surgery finished outside protocol window | 1 | 1
Not completed — Patient died outside SAE report period | 1 | 0
Not completed — Patient did not attend scheduled visit | 2 | 1
Not completed — Patient did not have surgery | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat Efficacy (ITT-E) population included all randomized participants who had received any study product, underwent the intended surgical procedure, and had an INR > 1.3 prior to the infusion. Participants in the ITT-E population were analyzed 'as randomized'.
Groups:
- Beriplex® P/N: Beriplex® P/N: Intravenous infusion, dosage depending on baseline INR, amount of coagulation factor IX and body-weight.
- Total: Total of all reporting groups
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma | Total
Number analyzed (Participants) | 87 | 81 | 168
Age, Customized [Number; unit: participants]
  < 65 years | 32 | 39 | 71
  >= 65 to < 75 years | 21 | 19 | 40
  >= 75 years | 34 | 23 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 31 | 68
  Male | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hemostatic Efficacy During Surgery
Description: Hemostatic efficacy was rated as excellent, good, or poor/none, based on prespecified definitions. Hemostatic efficacy was the binary endpoint of effective or non-effective hemostasis, where 'effective' was a hemostatic efficacy rating of "excellent" or "good," and 'non-effective' was a hemostatic efficacy rating of "poor/none".
Time Frame: From the start of infusion until the end of surgery
Population: The Intention-to-Treat Efficacy ITT-E population included all randomized participants who had received any study product, underwent the intended surgical procedure, and had an INR > 1.3 prior to the infusion. Participants in the ITT-E population were analyzed 'as randomized'.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 87 | 81
percentage of participants | 89.7 [83.3 to 96.1] | 75.3 [65.9 to 84.7]
Statistical Analysis 1: Comparison: Beriplex® P/N vs Fresh Frozen Plasma; The analysis of hemostatic efficacy was via calculation of the 95% confidence interval (CI) for the difference (Beriplex minus plasma) in the percentage of participants with effective hemostasis; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was -(minus)10%. If the lower limit of the 2-sided 95% CI was >-10%, then the null-hypothesis was rejected and it was concluded that Beriplex was non-inferior to plasma. The sample size estimation assumed that hemostatic efficacy would be rated 'effective' in 85% of participants in the plasma group and 90% of participants in the Beriplex group. The power to show non-inferiority with these assumptions was greater than 80% for two treatment groups of 80 participants; 95% confidence interval — No P-value is provided as non-inferiority was assessed via calculation of the 95% CI for the difference (Beriplex minus plasma) in the percentage of participants with effective hemostasis; The Newcombe-Wilson score method was used to estimate the 95% CI for the difference (Beriplex-plasma) in the % participants with effective hemostasis; Difference in effective hemostasis (%) = 14.3, 95% CI 2-sided [2.8 to 25.8]

2. Primary Outcome: Percentage of Participants Who Had a Rapid Decrease of the INR
Description: A rapid decrease of the INR was defined as an INR ≤ 1.3 at 30 minutes after the end of infusion. The INR is a standard way to describe the time it takes for blood to clot; an INR range of 0.8 to 1.2 is considered normal for a healthy person who is not using oral anticoagulant therapy.
Time Frame: 30 minutes after the end of infusion
Population: The ITT-E population included all randomized participants who had received any study product, underwent the intended surgical procedure, and had an international normalized ratio INR > 1.3 prior to the infusion. Participants in the ITT-E population were analyzed 'as randomized'.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 87 | 81
percentage of participants | 55.2 [44.7 to 65.6] | 9.9 [3.4 to 16.4]
Statistical Analysis 1: Comparison: Beriplex® P/N vs Fresh Frozen Plasma; The analysis of rapid decrease of the INR was via calculation of the 95% CI for the difference (Beriplex minus plasma) in the percentage of participants with INR ≤ 1.3 at 30 minutes after the end of infusion; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Newcombe-Wilson score method — [p-value comment as in outcome 1, analysis 1]; The Newcombe-Wilson score method was used to estimate the 95% CI for the difference (Beriplex-plasma) in the % pts with rapid decrease of the INR; Difference in effective hemostasis (%) = 45.3, 95% CI 2-sided [31.9 to 56.4]

3. Secondary Outcome: Plasma Levels of Factors II, VII, IX, and X, Protein C, and Protein S
Description: Plasma levels are presented as the percentage of normal at pre-infusion and 30 min and 24 h after the start of infusion. The plasma level assay results are reported as a potency relative to a standard, where 100% is considered to be normal.
Time Frame: From pre-infusion until 24 h after the start of infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of normal
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 85 | 79
percentage of normal
  Factor II, pre-infusion (n = 85; 79) | 32.0 (19.93) | 34.8 (26.19)
  Factor II, 0.5 h after infusion start (n = 71; 73) | 84.5 (20.92) | 42.5 (25.71)
  Factor II, 24 h after infusion start (n = 81; 74) | 81.4 (24.83) | 65.6 (23.68)
  Factor VII, pre-infusion start (n = 85; 79) | 36.8 (59.27) | 31.1 (25.16)
  Factor VII, 0.5h after infusion start (n = 71; 73) | 60.1 (44.91) | 41.6 (42.90)
  Factor VII, 24 h after infusion start (n = 81; 74) | 85.5 (59.76) | 83.7 (58.90)
  Factor IX, pre-infusion (n = 85; 79) | 48.1 (25.62) | 55.8 (30.50)
  Factor IX, 0.5 h after infusion start (n = 71; 73) | 71.6 (25.38) | 56.2 (23.12)
  Factor IX, 24 h after infusion start (n = 81; 74) | 85.2 (33.39) | 93.7 (34.25)
  Factor X, pre-infusion (n = 85; 79) | 19.3 (19.32) | 20.8 (21.38)
  Factor X, 0.5 h after infusion start (n = 71; 73) | 82.3 (23.33) | 29.8 (22.51)
  Factor X, 24 h after infusion start (n = 81; 74) | 78.3 (25.62) | 60.2 (22.44)
  Protein C, pre-infusion (n = 85; 78) | 48.8 (19.07) | 47.6 (21.38)
  Protein C, 0.5 h after infusion start (n = 71; 73) | 97.1 (21.97) | 52.5 (18.69)
  Protein C, 24 h after infusion start (n = 81; 74) | 87.3 (26.28) | 78.1 (24.80)
  Protein S, pre-infusion (n = 85; 79) | 45.25 (18.498) | 46.18 (20.986)
  Protein S, 0.5 h after infusion start (n = 72; 73) | 80.73 (31.489) | 55.82 (24.689)
  Protein S, 24 h after infusion start (n = 82; 74) | 75.97 (36.449) | 69.32 (27.504)

4. Secondary Outcome: Transfusion of Packed Red Blood Cells (PRBCs) or Whole Blood
Description: The total units of transfused PRBCs or whole blood
Time Frame: From the start of surgery until 24 h after the start of surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units of PRBCs or whole blood
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 87 | 81
units of PRBCs or whole blood | 0.3 (0.90) | 0.4 (1.02)

5. Secondary Outcome: Percentage of Participants With INR Correction at Various Times After the Start of Infusion
Description: The time taken from the start of infusion to INR correction (defined as an INR ≤ 1.3) was recorded. The percentage of participants with INR correction was calculated at 0.5, 1, 3, 6, 12, and 24 h after the start of infusion.
Time Frame: From the start of infusion until INR correction; calculated at 0.5, 1, 3, 6, 12, and 24 h after the start of infusion
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 87 | 81
percentage of participants
  0.5 h | 1 | 0
  1 h | 54 | 0
  3 h | 77 | 10
  6 h | 81 | 20
  12 h | 83 | 32
  24 h | 87 | 48

6. Secondary Outcome: Percentage of Participants Who Received Red Blood Cells
Description: Red blood cells were PRBCs and whole blood
Time Frame: From the start of surgery until 24 h after the start of surgery
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 87 | 81
percentage of participants | 16.1 | 14.8

7. Secondary Outcome: Overall Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs. TEAEs were defined as adverse events that developed or worsened following exposure to investigational medicinal product. Treatment-related TEAEs were events whose relationship to study treatment was related, probably related, or possibly related in the opinion of the investigator. Treatment emergent adverse events with missing relationship were considered related to treatment. Serious TEAEs were treatment-emergent serious adverse events (SAEs).
Time Frame: From the start of infusion up to the allowed time window of the Day 10 visit for non-serious AEs and from the start of infusion up to the allowed time window of the Day 45 visit for SAEs
Population: The Intention-to-Treat Safety (ITT-S) population included all participants who were randomized and who had received any portion of study product. Participants in the ITT-S population were analyzed 'as treated'.
Measure: Number; unit: participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 88 | 88
participants
  Any TEAE | 49 | 53
  At least possibly treatment-related TEAE | 8 | 15
  Serious TEAE | 22 | 23
  Death | 4 | 8

ADVERSE EVENTS:
Time Frame: From the start of infusion up to the allowed time window of the Day 10 visit for non-serious AEs and from the start of infusion up to the allowed time window of the Day 45 visit for SAEs.
Description: The AEs presented were serious and non-serious (other) TEAEs. The ITT-S population included all subjects who were randomized and who had received any portion of study product. Participants in the ITT-S population were analyzed 'as treated'. "General disorders" were collected under the MedDRA SOC General disorders and administration site conditions.
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Serious Adverse Events (participants affected / at risk) | 22/88 | 23/88
Other Adverse Events (participants affected / at risk) | 41/88 | 44/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beriplex® P/N (N=88) | Fresh Frozen Plasma (N=88)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Wound necrosis (General disorders) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beriplex® P/N (N=88) | Fresh Frozen Plasma (N=88)
Constipation (Gastrointestinal disorders) | 10 (10) | 4 (4)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 8 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (6) | 3 (3)
Tachycardia (Cardiac disorders) | 5 (5) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 6 (6) | 6 (6)
Pyrexia (General disorders) | 3 (3) | 5 (5)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Confusional state (Psychiatric disorders) | 3 (4) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 6 (6)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 3 (3)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Body temperature increased (Investigations) | 3 (3) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.